CLINICAL TRIAL: NCT00823420
Title: Influence of a Prematuration Culture With a PDE3-I on Embryonic Aneuploidy Rate and Developmental Potential
Brief Title: Influence of a Prematuration Culture With a Phosphodiesterase-3 Inhibitor (PDE3-I) on Embryonic Aneuploidy Rate and Developmental Potential
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Prematuration Culture With a Phosphodiesterase-3 Inhibitor (PDE3-I) has been replaced by a different formulation
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: University of Adelaide (Other); Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IWT-JSMDV2008
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2009-01

CONDITIONS: Infertility
Keywords: PCOS and normal ovulatory patients; aneuploidy; in-vitro maturation of oocytes
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome; Aneuploidy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- in-vitro maturation of oocytes (Experimental)
  Interventions: Procedure: prematuration culture

INTERVENTIONS:
Procedure: prematuration culture — The aneuploidy rate and the developmental potential of embryos obtained from PDE3 inhibitor-treated oocytes (a "prolonged" IVM (PMC)) in comparison to "conventional" IVM will be analysed. It is intended to assess the nuclear and cytogenetic constitution of the obtained embryos.

SUMMARY:
A single centre randomised controlled trial investigating the influence of a novel prematuration system (PMS) using a phosphodiesterase-3 inhibitor for in-vitro maturation of oocytes

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers, either with PCOS/PCOS-like ovaries, or with normal ovaries, who undergo oocyte donation for research
* AFC at least 10
* AMH: > 5 μg/L
* Female age < 36 years

Exclusion Criteria:

* major uterine or ovarian abnormalities

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2009-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of aneuploidy rate by fluorescence in situ hybridisation (FISH) technique in 6 to 8 cell embryos from prolonged (PMC) IVM compared to conventional IVM on sibling oocytes. | 3 days after egg retrieval

SECONDARY OUTCOMES:
Implantation potential of embryos from conventional IVM performed on Type II COC. Efficiency of both maturation systems in obtaining blastocysts. Endometrium quality in IVM cycles. | 7 days after egg retrieval

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Reproductive Medicine, Brussels, Belgium